CLINICAL TRIAL: NCT01096654
Title: Towards Cost-effective Management of Patients With Hypertension Due to Primary Aldosteronism: Adrenal Vein Sampling or Ct-scan?
Brief Title: SPARTACUS: Subtyping Primary Aldosteronism: a Randomized Trial Comparing Adrenal Vein Sampling and Computed Tomography Scan.
Acronym: SPARTACUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: avs-ct1
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Hyperaldosteronism
Keywords: endocrine hypertension; primary hyperaldosteronism; aldosterone; aldosterone-producing adenoma; bilateral adrenal hyperplasia; computed tomography; adrenal vein sampling
MeSH Terms: conditions — Hyperaldosteronism; Adrenocortical Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CT-scan (Active Comparator): In this group treatment will be based on the outcome of the CT-scan only. Patients will be treated by adrenalectomy (Adx) if an unilateral lesion is visible on the CT-scan and the contralateral gland is normal. If bilateral lesions, bilateral enlargement or symmetric normal adrenal glands are present patients will be treated by the mineralocorticoid receptor antagonist (MRA)
  Interventions: Other: Ct-scan or adrenal vein sampling
- Adrenal Vein Sampling (Active Comparator): This group will be treated according to the results of the adrenal vein sampling only. Adrenal vein sampling will be performed under the continuous infusion of ACTH (adrenocorticotropic hormone). A cortisol ratio ≥ 3 between the adrenal vein and the inferior vena cava is set as the criterium for successful cannulation. The criterium for lateralization is a aldosterone/cortisol ratio ≥ 4 between the adrenal veins and a lower aldosterone/cortisol ratio in the contralateral adrenal vein than in the inferior vena cava.
  If AVS fails patients will be treated according to the CT-findings as described in the group with CT-scan only. Patients with a successful AVS will be treated by Adrenalectomy if unilateral production of aldosterone is shown. If no unilateral aldosterone production is present, i.e. the aldosterone/cortisol ratio is less than 4, patients will be treated by MRA.
  Interventions: Other: Ct-scan or adrenal vein sampling

INTERVENTIONS:
Other: Ct-scan or adrenal vein sampling — Patients will be randomized to undergo either adrenal CT-scanning or AVS (with pre-AVS adrenal CT-scanning for phlebography). The result of either of these tests will determine the course of action: adrenalectomy for adenoma or MRAs for bilateral hyperplasia.

SUMMARY:
Rationale: Primary hyperaldosteronism (PA) is the most frequent form of secondary hypertension. In PA autonomous hypersecretion of aldosterone by one or both adrenal glands causes hypertension that is often refractory to treatment. PA is usually caused by either a unilateral aldosterone-producing (micro)adenoma (APA) or by bilateral adrenal hyperplasia (BAH). Distinction between APA and BAH is critical since the former is treated with the aim of cure by adrenalectomy, and the latter by mineralocorticoid receptor antagonists. This distinction can be made by adrenal vein sampling (AVS), as recommended by The Endocrine Society 2008 guideline or by CT-scanning, as is common practice in the Netherlands. AVS is invasive, demands great skill, and is expensive, while CT-scanning is non-invasive, easy and cheap, but might be less accurate. However, the advantage of AVS has never been demonstrated in prospective randomized studies. Here we propose to perform a prospective, randomized, multicenter study that compares effectiveness of AVS with effectiveness of CT-scanning for the diagnosis of PA subtype.

Objective: To assess the quantity of antihypertensive medication needed in order to normalize blood pressure in patients who have been managed for PA according to either AVS or CT-scan. Secondary objectives: to assess potassium, costs of management and quality of life.

Study design: Prospective, randomized trial in a multi-centre setting. Two hundred patients will be recruited within two years. Follow-up will be one year after (start of) treatment.

Study population: Adult patients with therapy-resistant hypertension, with or without hypokalemia, caused by PA.

Intervention: Patients will be randomized to undergo either adrenal CT-scanning or AVS (with pre-AVS adrenal CT-scanning for phlebography). The result of either of these tests will determine the course of action: adrenalectomy for adenoma or MRAs for bilateral hyperplasia.

Main study parameters/endpoints: The quantity of antihypertensive drugs patients are using to obtain target blood pressure, expressed in Daily Defined Dosages, is used as the main study parameter. There is no criterion standard for accuracy of the diagnosis of PA-subtype, but we assume that if treatment is based on a more accurate diagnosis, treatment is more effective. The most important secondary endpoints are the costs of the diagnostic course and long-term medical treatment and the quality of life as assessed by a validated questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Legally capacitated;
* ≥ 18 years of age;
* Diagnosed with hypertension that is difficult to treat (blood pressure > 140/90 mmHg in spite of two antihypertensive drugs in adequate doses), or accompanied by hypokalemia, either spontaneous or induced by use of diuretics;
* patients must have a positive result on a sodium loading test (as recommended in the Endocrine Society Guideline), i.e. insufficient suppression of aldosterone.
* Cooperating patient who is willing to undergo adrenal surgery in case of an adenoma or lateralized aldosterone secretion, who is able to comply with the study protocol and who is willing to give written informed consent.

Exclusion Criteria:

* Unsuitability for or objection to undergo AVS, CT or adrenal surgery.(including pregnancy);
* Glucocorticoid remediable aldosteronism or adrenal carcinoma;
* Severe or terminal co-morbidity which seriously interferes with possible treatment or health related quality of life;
* Requirement of certain medication that interacts with the prescribed treatments in this protocol or that can cause hypertension as an important side-effect e.g. glucocorticoids. Patients will only be excluded as the medication cannot be stopped or altered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Daily Defined Doses of antihypertensive medication | assessed after 1 year of follow-up
  The main study parameter is the quantity of antihypertensive drugs patients are using to obtain target blood pressure, expressed in Daily Defined Doses (DDD)16. The DDD is the assumed average maintenance dose per day for a drug used for its main indication in adults. It provides a fixed unit of measurement independent of price and dosage form (e.g. tablet strength) enabling the researcher to assess trends in drug consumption and to perform comparisons between population groups.

SECONDARY OUTCOMES:
Total cost of diagnosis and management | assessed after 1 year follow-up
  Costs of the diagnostic course and the first year of treatment after determination of subtype of PA will be calculated prospectively and bottom-up for each participant. This includes costs of CT, AVS (hardware, rent of facility, lab determinations, cost of personnel), operation, outpatient clinic visits, medication and lab controls for potassium and creatinine. Long term costs will be extrapolated from the first year's results for an average life expectancy and a predefined discounting rate.
Health Related Quality of Life | assesed before treatment, at 6 months and at 12 months follow-up
  The quality of life in our patients may be influenced in different ways. AVS is more invasive and more burdensome to the patient than CT; the same holds for surgery as compared to medical treatment; on the other hand, more intense and prolonged (lifelong) antihypertensive drug treatment may be associated with more side effects. We suggested to explore these issues, using the . EQ-5D (European Quality of Life-5 Dimensions) and the SF-36 (Medical Outcomes Study 36-Item Short-Form Health Survey). This will allow for a detailed analysis of the impact of the two strategies on the quality of life of the patients.
Potassium level | assesed before treatment and after 1 year follow-up
  Serum potassium levels will be determined before Adx or start of MRA and one year later. Potassium levels will be compared between the two arms of the study.
Result of a sodium loading test | assessed after 1 year follow-up
  This test, which is the reference test for the existence of PA, will be performed only in patients that have undergone adrenalectomy because in these patients PA is expected to be cured after adrenalectomy with hence a normal result of this test. The test will be performed 1 year after operation after interruption of medication that interferes with the measurement of aldosterone levels. The proportion of patients who were cured (i.e. with normal saline loading test) will be compared between the CT- and the AVS-group.
Post-hoc analysis: medication dosage | assessed after 1 year follow-up
  A post-hoc analysis on medication use will be performed using different outcome measures. Required antihypertensive medication one year after the (start of) treatment, expressed in multiples of the recommended starting dose and fraction of the recommended maximum dose, will be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Deinum, Dr., Principal Investigator — UCM St. Radboud
Locations (1):
- UMC St. radboud, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Kempers MJ, Lenders JW, van Outheusden L, van der Wilt GJ, Schultze Kool LJ, Hermus AR, Deinum J. Systematic review: diagnostic procedures to differentiate unilateral from bilateral adrenal abnormality in primary aldosteronism. Ann Intern Med. 2009 Sep 1;151(5):329-37. doi: 10.7326/0003-4819-151-5-200909010-00007. PMID 19721021
- [Background] Mulatero P, Bertello C, Sukor N, Gordon R, Rossato D, Daunt N, Leggett D, Mengozzi G, Veglio F, Stowasser M. Impact of different diagnostic criteria during adrenal vein sampling on reproducibility of subtype diagnosis in patients with primary aldosteronism. Hypertension. 2010 Mar;55(3):667-73. doi: 10.1161/HYPERTENSIONAHA.109.146613. Epub 2010 Feb 1. PMID 20124107
- [Background] Kline GA, Harvey A, Jones C, Hill MH, So B, Scott-Douglas N, Pasieka JL. Adrenal vein sampling may not be a gold-standard diagnostic test in primary aldosteronism: final diagnosis depends upon which interpretation rule is used. Variable interpretation of adrenal vein sampling. Int Urol Nephrol. 2008;40(4):1035-43. doi: 10.1007/s11255-008-9441-9. Epub 2008 Aug 12. PMID 18696249
- [Background] Stewart PM, Allolio B. Adrenal vein sampling for Primary Aldosteronism: time for a reality check. Clin Endocrinol (Oxf). 2010 Feb;72(2):146-8. doi: 10.1111/j.1365-2265.2009.03714.x. Epub 2009 Sep 21. No abstract available. PMID 19769616
- [Derived] Velema M, Dekkers T, Hermus A, Timmers H, Lenders J, Groenewoud H, Schultze Kool L, Langenhuijsen J, Prejbisz A, van der Wilt GJ, Deinum J; SPARTACUS investigators. Quality of Life in Primary Aldosteronism: A Comparative Effectiveness Study of Adrenalectomy and Medical Treatment. J Clin Endocrinol Metab. 2018 Jan 1;103(1):16-24. doi: 10.1210/jc.2017-01442. PMID 29099925
- [Derived] Dekkers T, Prejbisz A, Kool LJS, Groenewoud HJMM, Velema M, Spiering W, Kolodziejczyk-Kruk S, Arntz M, Kadziela J, Langenhuijsen JF, Kerstens MN, van den Meiracker AH, van den Born BJ, Sweep FCGJ, Hermus ARMM, Januszewicz A, Ligthart-Naber AF, Makai P, van der Wilt GJ, Lenders JWM, Deinum J; SPARTACUS Investigators. Adrenal vein sampling versus CT scan to determine treatment in primary aldosteronism: an outcome-based randomised diagnostic trial. Lancet Diabetes Endocrinol. 2016 Sep;4(9):739-746. doi: 10.1016/S2213-8587(16)30100-0. Epub 2016 Jun 17. PMID 27325147